CLINICAL TRIAL: NCT05902468
Title: A Clinical Study Evaluating the Use od Ursodeoxycholic Acid as Adjuvant Therapy in Type 2 Diabetes Mellitus
Brief Title: Ursodeoxycholic Acid as add-on Therapy in Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Principal Investigator, Eman Ghonaim, Eman Mabrouk Mahmoud Ghonaim, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4/2023 INTM
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): 44 diabetic patients receiving dual treatment with metformin and dipeptidyl peptidase-4 (DPP-4) inhibitors (such as vildagliptin)
- Group 2 (Active Comparator): 44 diabetic patients who will receive ursodeoxycholic acid 500 mg orally twice daily in addition to dual treatment with metformin and dipeptidyl peptidase-4 (DPP-4) inhibitors (such as vildagliptin)
  Interventions: Drug: Ursodeoxycholic acid

INTERVENTIONS:
Drug: Ursodeoxycholic acid — ursodeoxycholic acid 500 mg orally twice daily for 12 weeks
  Arms: Group 2

SUMMARY:
Diabetes mellitus (DM) is a complex metabolic disorder characterized by hyperglycemia and abnormalities in carbohydrate, fat, and protein metabolism. It is one of the most prevalent metabolic disorders globally. Despite the advancement in anti-diabetic drug therapy, most patients fail to achieve optimal glycemic control. therefore, there is a large unmet need to develop new strategies to improve the therapeutic outcomes in diabetic patients. This study is designed to evaluate the efficacy of ursodeoxycholic acid as adjunctive therapy in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a complex metabolic disorder characterized by hyperglycemia and abnormalities in carbohydrate, fat, and protein metabolism. It is one of the most prevalent metabolic disorders globally. More than 75% of diabetic patients live in low- and middle-income countries. About 90% of diabetic patients have type 2 diabetes.

Insulin resistance (IR) and β-cell dysfunction are the two main pathophysiological events contributing to type 2 diabetes.

Insulin resistance is a pathological condition in which insulin-dependent tissues fail to properly respond to normal circulatory levels of insulin. Inflammatory mediators play a key role in insulin resistance. For example, tumor necrosis factor alpha (TNF-α) impairs insulin signaling via serine phosphorylation of insulin receptor substrate (IRS-1). Additionally, it reduces glucose transporter-4 (GLUT-4) expression, limiting glucose entry into adipocytes and skeletal muscle cells. Similarly, IL-6 induces IRS degradation. Oxidative stress interferes with insulin signal transduction leading to IR. It activates several serine-threonine kinase pathways, which, in turn, phosphorylates IRS proteins leading to subsequent degradation.

β-cell dysfunction is associated with β-cell death. In an excessive nutritional state, as in obesity, hyperglycemia and hyperlipidemia are often present, favoring IR and chronic inflammation. Under these circumstances, β-cells are subject to toxic pressures including inflammation, endoplasmic reticulum stress, oxidative stress, as well as amyloid stress, that ultimately lead to loss of islet integrity.

Ursodeoxycholic acid (UDCA) is an endogenous hydrophilic bile acid normally present in human bile and traditionally used for the treatment of liver diseases. UDCA has direct antioxidant properties. It decreased glucose levels, alleviated hyperinsulinemia, and improved islet function in rats with liver fibrosis. Therefore, this study is designed to evaluate the efficacy of ursodeoxycholic acid as adjunctive therapy in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with type 2 diabetes mellitus within the previous 12 months.
* Glycated hemoglobin (HbA1c) between 7% and 9%.
* Body mass index ≥ 25 kg/m2

Exclusion Criteria:

* Pregnant or nursing women.
* Type 1 diabetes mellitus.
* Liver disease (alanine aminotransferase > 3 upper normal limit).
* Kidney disease (estimated glomerular filtration rate < 60 ml/min/1.73 m2).
* Inflammatory bowel diseases
* History of allergy and/or adverse reactions to the drugs used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-06-28 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-11-28 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | 12 weeks
  Fasting blood glucose, glycated hemoglobin

SECONDARY OUTCOMES:
Lipid profile | 12 weeks
  Total cholesterol, triglycerides, HDL-cholesterol, and LDL-cholesterol
Insulin resistance | 12 weeks
  Fasting insulin, HOMA-IR
Oxidative stress marker | 12 weeks
  Serum malondialdehyde
Inflammation marker | 12 weeks
  Interleukin-6, high mobility group box-1
Serum asprosin | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of medicine, Tanta University, Tanta, El-Gharbia
  - Faculty of Medicine, Menoufia University, Shibīn al Kawm, Menoufia